CLINICAL TRIAL: NCT03055702
Title: Using Mobile Phone Short Message Service (SMS) Reminders to Enhance Type 2 Diabetes Mellitus Appointment Attendance in a Primary Care Clinic
Brief Title: Using Mobile Phone Short Message Service (SMS) Reminders to Enhance Appointment Attendance in DM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KW/EX-16-104(100-10)
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Appointments and Schedules; Diabetes Mellitus, Type 2
Keywords: Short Message Service; appointment reminder; Attendance rate
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS group (Experimental): receive a mobile phone text reminder for scheduled clinic appointment 24-72 hours before,
  Interventions: Other: Mobile phone text message reminder
- Usual care group (No Intervention): Usual care, either telephone reminder or no reminder

INTERVENTIONS:
Other: Mobile phone text message reminder — an SMS remind subjects to come for scheduled clinic appointment 24-72 hours before
  Arms: SMS group

SUMMARY:
A randomized controlled trial of patients with type 2 diabetes mellitus with multiple appointments into short message service group and control group. The attendance rate of these two groups of patients will be compared.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the appointment attendance rate using SMS reminder of nurses and allied health appointments for diabetic patients, when compared to conventional telephone reminder and no reminder. We also aim at determine the factors associated with appointment attendance. Finally, we will also survey patients' acceptance and satisfaction to the SMS service.

This is a single blind randomization study. It will be carried out in Ha Kwai Chung General Outpatient Clinic.

The primary outcome of this study is to evaluate the attendance rate of each individual doctor, nurses and allied health clinic appointments for diabetic patients, as well as their overall attendance rates:

1. Diabetes Complication Screening Clinic (OPAS DMCS/RDNA)
2. Diabetes Nurse Intervention Clinic (OPAS DMIC/RDNI)
3. DM nurse group (OPAS RDNG)
4. Dietitian Counselling (OPAS DC/DG)
5. Physiotherapy (OPAS PTC/PTG)
6. Diabetes Doctor Session (OPAS RDR)
7. Retino photo Assessment (OPAS RDO)
8. Blood taking appointment (OPAS LABT)

The secondary outcomes are:

* Acceptance Rate of SMS Reminder Vs Telephone Reminder Vs no reminder
* Factors associated with acceptance of SMS

  1. Personal Parameters: Age, sex, educational level, occupation, mobile phone models, Habit of using mobile phone service
  2. Disease Parameters: Number and types of comorbidity, disease control (by biochemical markers)
  3. Quality of Life (by SF-6D)
* Reported adverse effects of the reminder system
* Chang in biochemical markers (BMI, HbA1c, LDL-c level) 6-9 months later

Subjects who agreed to participate in this study will first receive a survey on the acceptance of SMS service. For those agree to receive SMS reminder, they will be randomized to:

1. an SMS remind them to come for scheduled clinic appointment 24-72 hours before, or
2. usual care with no reminder / telephone reminder.

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of type 2 diabetes
* Have more than 1 clinic services appointment under RAMP-DM programme:

  (e.g. blood taking, diabetic nurse individual counselling, group education, diabetic complication screening, retinal photo assessment, dietician counselling, etc)

Exclusion Criteria:

1. Cannot read or receive appointment schedule on mobile phone
2. Do not speak Cantonese/English or read Chinese/English
3. Mentally incapacitated
4. Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Attendance Rate of the scheduled clinic appointment | between booking time and appointment time, usually within 1 weeks to 16 weeks
  Attendance Rate

CONTACTS AND LOCATIONS:
Overall Officials: Man Chi Dao, M.B.B.S., Principal Investigator — Resident
Locations (1):
- Ha Kwai Chung General Outpatient Clinic, Kwai Chung, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided